CLINICAL TRIAL: NCT00319215
Title: A Study to Investigate the Residual Effects of Ramelteon (8 mg), Zopiclone (7.5 mg) and Placebo on Actual Driving, Memory, Psychomotor Performance and Mood
Brief Title: Effects of Ramelteon on Driving Ability
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Utrecht Institute for Pharmaceutical Sciences (Other)
Collaborators: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 05/316; Studynumber:TAK-375/EC103; EudraCT Number 2005-005553-22
Record Dates: First submitted 2006-04-26; First posted 2006-04-27 (Estimated); Last update posted 2007-04-25 (Estimated); Status verified 2007-04

CONDITIONS: Insomnia
Keywords: ramelteon; zopiclone; driving; memory; balance; psychomotor
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — ramelteon; zopiclone

INTERVENTIONS:
Drug: Ramelteon 8 mg
Drug: Zopiclone 7.5 mg

SUMMARY:
The primary purpose of this study is to investigate the effects of bedtime administration of a single dose of ramelteon (8 mg), zopiclone (7.5 mg), and placebo on next-morning on-road driving performance. In addition, the drugs' effects on balance are evaluated during the night, and the next morning residual effects on memory and psychomotor performance.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is male or female, 21 - 55 years of age, inclusive
2. The subject is capable of understanding and complying with the protocol requirements.
3. The subject or the subject's legally acceptable representative signs a written, informed consent form prior to the initiation of any study procedures.
4. The subject, if female, is non-pregnant and non-lactating.
5. Possession of a valid driver's license for at least 3 years and a reported history of having driven at least 5000 km per year on average, for the last 3 years prior to entering into the trial.
6. An SDLP level at the end of the driving test of the dress rehearsal that does not exceed 24 cm. This dress rehearsal is performed at Visit 1.

Exclusion Criteria:

1. The subject has a known hypersensitivity to ramelteon, zopiclone or related compounds, including melatonin.
2. The subject has participated in any other investigational study and/or taken any investigational drug within 30 days or five half-lives prior to the first night of double-blind study medication, whichever is longer.

5.History or presence of any clinically significant gastrointestinal, cardiovascular, hepatic, renal, haematological, endocrine, respiratory, neurological or psychiatric disease 6.History of primary insomnia (DSM IV-TR criteria) within the past 6 months. 7.The subject has used any medication with psychotropic effects (e.g. antidepressants, anxiolytics, antihistamines) within 30 days of the initial visit.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30
Dates: Start 2006-03; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Standard Deviation of Lateral Position (SDLP); i.e. the weaving of the car.
Standard Deviation of Speed (SDS)

SECONDARY OUTCOMES:
Mean Speed (MS)
Mean Lateral Position (MLP)
Word Learning test:Immediate recall, Delayed Recall, Recognition time & score
Sternberg memory scanning test: reaction time and % errors
Tracking task: RMS (tracking error)
Divided attention test: RMS,reaction time and % errors
DSST: number of copied symbols

CONTACTS AND LOCATIONS:
Overall Officials: Joris Verster, PhD, Principal Investigator — Utrecht Institute for Pharmaceutical Sciences
Locations (1):
- Utrecht Institute for Pharmaceutical Sciences, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Mets MA, de Vries JM, de Senerpont Domis LM, Volkerts ER, Olivier B, Verster JC. Next-day effects of ramelteon (8 mg), zopiclone (7.5 mg), and placebo on highway driving performance, memory functioning, psychomotor performance, and mood in healthy adult subjects. Sleep. 2011 Oct 1;34(10):1327-34. doi: 10.5665/SLEEP.1272. PMID 21966064